CLINICAL TRIAL: NCT02496728
Title: American Heart Association Strategically Focused Research Network: mHealth Intervention to Preserve and Promote Ideal Cardiovascular Health
Brief Title: NUYou:mHealth Intervention to Preserve and Promote Ideal Cardiovascular Health
Acronym: NUYou
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Bonnie Spring, Professor Preventive Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14SFRN20480260
Record Dates: First submitted 2015-05-29; First posted 2015-07-14 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Cardiovascular Disease
Keywords: Mobile Health; Smartphone; Cardiovascular health; College students; Smoking; Physical activity; Diet; BMI; Blood pressure; Cholesterol; Glucose; Text; Facebook; Instagram; Push Notifications; Ecological Momentary Assessment
MeSH Terms: conditions — Cardiovascular Diseases; Smoking; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardiovascular Health (Experimental): Participants will be given the results of their health assessment and feedback regarding their health behaviors and overall health. Recommendations for change will be given if warranted. Participants will download the study's mobile health application on their smartphone. They will then be asked to report once a week about their health behaviors on the application. Participants will also be asked to self-monitor health behaviors that are not already at ideal levels using the study application (environmental cues). Participants will be asked to join a secret Facebook group where informational materials will be posted, participants can post about study health behaviors and social interaction around health behaviors can occur (social support and environmental cues).
  Interventions: Behavioral: Mobile Health Application; Behavioral: Environmental Cues; Behavioral: Social Support; Behavioral: Educational Materials
- Whole Health (Active Comparator): Participants will be given the results of their health assessment. They will then receive educational materials about sunscreen use, safe sex, hydration and vehicular safety. Participants will download the study's mobile health application on their smartphone. They will then be asked to report once a week about their health behaviors on the application. Participants will also be asked to self-monitor how much water they drink using the study application. Participants will be asked to join a secret Facebook group where informational materials will be posted, they can post about study health behaviors and social interaction around health behaviors can occur (social support and environmental cues).
  Interventions: Behavioral: Mobile Health Application; Behavioral: Environmental Cues; Behavioral: Social Support; Behavioral: Educational Materials

INTERVENTIONS:
Behavioral: Mobile Health Application — An application on a smart phone that is designed to help individuals self-monitor health behaviors.
Behavioral: Environmental Cues — Text messages, informational posts and reminders supporting healthy behaviors.
Behavioral: Social Support — Participants may interact with each other through a private Facebook group.
Behavioral: Educational Materials — Educational materials regarding healthy behaviors.

SUMMARY:
The purpose of the study is to investigate the preservation or promotion of health in students during the college years.

DETAILED DESCRIPTION:
Freshman college students at Northwestern University will be cluster randomized to two groups based on their dorm. The intervention for one group will target smoking, physical activity, BMI and consumption of fruits and vegetables. The intervention in the second group will target traveling behavior, sexual risk behaviors, sunscreen use and hydration. Baseline health and lifestyle measures will be assessed for each participant prior to intervention. Health assessments will measure height, weight, fasting glucose, total cholesterol and carbon monoxide. The lifestyle measure will ask questions about physical activity, diet, alcohol and tobacco use, safe sex practices, driving habits, and sunscreen use. These same measures will be repeated during the fall of the students' sophomore and junior years.

Participants will be given a mobile application and encouraged to track some behaviors. In addition, participants will be asked to answer weekly questions regarding health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Freshman at Northwestern University in the fall of 2015
* Live on campus
* Read, write and speak English
* Own an Iphone or Android smart phone

Exclusion Criteria:

* Pregnant or trying to become pregnant
* Established cardiovascular disease
* Unstable psychiatric or medical condition

Ages: 17 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 302 (Actual)
Dates: Start 2015-05; Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
American Heart Association MyLifeCheck (Simple 7) score as a measure of cardiovascular health | 2 years
  Participant's Simple 7 score is the sum of 7 cardiovascular health metrics attained at ideal levels as defined by American Heart Association. 1) physically active - Exercising at least 150 minutes of moderate or 75 minutes of vigorous physical activity per week. 2) Good diet quality - Eating 5 servings of fruits and vegetables per day, at least 3 servings of whole grain, and no more than 16 oz. of soda per day, rarely or never eats high sodium foods or processed meats. 3) nonsmoking - nonsmoker for at least a year. 4) not overweight - BMI < 25 kg/m2. 5) normoglycemic - fasting glucose < 100 mg/dl. 6) not hypercholesterolemic : total Cholesterol < 200 mg/dl. 7) not hypertensive. Blood Pressure <120/<80.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Spring, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pfammatter AF, Champion KE, Finch LE, Siddique J, Hedeker D, Spring B. A mHealth intervention to preserve and promote ideal cardiovascular health in college students: Design and protocol of a cluster randomized controlled trial. Contemp Clin Trials. 2020 Nov;98:106162. doi: 10.1016/j.cct.2020.106162. Epub 2020 Oct 8. PMID 33038506